CLINICAL TRIAL: NCT02099708
Title: Takepron Capsules 15/ Orally Dispersing（OD） Tablets 15 Special Drug Use Surveillance Long-term Use Survey on the Prevention of Recurrence of Gastric/Duodenal Ulcer in Patients Receiving Non-steroidal Anti-inflammatory Drugs
Brief Title: Long-term Use of Takepron on the Prevention of Recurrence of Gastric/Duodenal Ulcer in Patients Receiving Non-steroidal Anti-inflammatory Drugs
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 467-713; JapicCTI-142418 (Registry Identifier: Japic CTI); JapicCTI-R150705 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-09

CONDITIONS: Gastric or Duodenal Ulcers
Keywords: Pharmacological therapy
MeSH Terms: conditions — Duodenal Ulcer | interventions — Lansoprazole; Tablets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lansoprazole 15 mg: Lansoprazole 15 mg, capsules or orally disintegrating (OD) tablets, orally, once, daily for up to 12 months.
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole Capsules 15 mg/ Orally Disintegrating (OD) Tablets 15 mg
  Other Names: Takepron Capsules 15 mg, Takepron Orally Disintegrating (OD) Tablets 15 mg

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of long-term administration of lansoprazole (Takepron) therapy for up to 12 months in the routine clinical setting in patients receiving oral non-steroidal anti-inflammatory drugs (NSAIDs)

DETAILED DESCRIPTION:
This is a special survey on long-term use (for up to 12 months) of lansoprazole (Takepron) to determine the incidence of adverse drug reactions in the routine clinical setting in patients receiving non-steroidal anti-inflammatory drugs (NSAIDs).

The usual adult dosage is 15 mg of lansoprazole administered orally once daily.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients with a history of gastric or duodenal ulcers (2) Patients requiring long-term use of NSAIDs for reasons such as pain management for rheumatoid arthritis or osteoarthritis (3) Patients taking oral NSAIDs at the start of administration of lansoprazole (including patients who start NSAIDs on the same day as the start of administration of lansoprazole)

Exclusion Criteria:

* (1) Patients with gastric or duodenal ulcer (in the active [A1, A2] or healing [H1, H2] stage if assessed endoscopically) at the start of administration of lansoprazole (2) Patients with active upper gastrointestinal hemorrhage at the start of administration of lansoprazole (3) Patients with contraindications for lansoprazole

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gastric or duodenal ulcers
Sampling Method: Non-Probability Sample
Enrollment: 3502 (Actual)
Dates: Start 2010-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 501 investigative sites in Japan from October 2010 to March 2014 (N=3,502).
Pre-assignment Details: Patients with a history of gastric or duodenal ulcers and requiring long-term use of nonsteroidal anti-inflammatory drugs were enrolled in the study.
Period: Overall Study
Arm/Group | Lansoprazole 15 mg
Started | 3502 (Number of cases.)
Safety Analysis Set (SAS) | 3302 (All participants who took the study drug at least once.)
Completed | 3302
Not Completed | 200
Not completed — Data Not Available | 30
Not completed — Lost to Follow-up | 141
Not completed — Other | 29

BASELINE CHARACTERISTICS:
Population: Safety analysis set: all participants who took the study drug at least once.
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3302
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2268
  Male | 1034
Purpose of Non-steroidal Anti-Inflammatory Drug (NSAID) Treatment [Number; unit: participants] — Participants could be counted in more than 1 category (including duplicates).
  participants
    Rheumatoid arthritis | 573
    Osteoarthritis | 1729
    Other | 1116
Details of the History of Gastric or Duodenal Ulcers: Site of Disease [Number; unit: participants] — Participants could be counted in more than 1 category (including duplicates).
  participants
    Gastric ulcer | 2632
    Gastroduodenal ulcer | 207
    Unknown | 490
Details of the History of Gastric or Duodenal Ulcers: Time of Emergence [Number; unit: participants]
  <6 months before treatment | 161
  ≥ 6 months to < 1 year before treatment | 63
  ≥ 1 year before treatment | 449
  Unknown | 2629
Presence or Absence of H. Pylori Infection [Number; unit: participants]
  Negative | 276
  Positive | 55
  Unknown | 2971

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Drug Reactions
Description: Frequency was defined as the number of participants for each adverse event Frequency, severity, and time to onset of adverse drug reactions tabulated by each symptom. Adverse events are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. Among these, events which are considered possibly associated with a medicinal product are defined as adverse drug reactions.
Time Frame: 12 months
Population: Safety analysis set (SAS) - All participants who received at least 1 dose of open-label study drug.
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3302
participants
  Bronchitis | 1
  Colon cancer | 1
  Depression | 1
  Cervical radiculopathy | 1
  Atrial fibrillation | 1
  Cardiac failure | 1
  Myocardial ischaemia | 1
  Abdominal discomfort | 4
  Abdominal pain upper | 1
  Colitis | 1
  Constipation | 2
  Diarrhoea | 8
  Enterocolitis | 1
  Nausea | 1
  Oral mucosal blistering | 1
  Stomatitis | 1
  Colitis microscopic | 1
  Faeces soft | 2
  Eczema | 1
  Hyperhidrosis | 1
  Rash | 1
  Generalised erythema | 1
  Osteoporosis | 2
  Feeling abnormal | 1
  Thirst | 2

2. Secondary Outcome: Presence or Absence of Endoscopic Examinations
Description: Summary of data on the presence or absence of gastric or duodenal ulcers by using endoscopic examinations.
Time Frame: From baseline to 12 months
Population: Efficacy Analysis Set: all participants from the SAS, excluding those for whom usage of NSAIDs during the treatment of lansoprazole was not confirmed and those who had gastric or duodenal ulcers at the start of administration of lansoprazole.
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3248
participants
  No | 3098
  Yes | 150

3. Secondary Outcome: Presence of Gastric or Duodenal Ulcer
Description: Summary of data on the presence or absence of gastric or duodenal ulcer.
Time Frame: From baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3248
Participants
  No | 3239
  Yes | 9

4. Secondary Outcome: Presence of Onset of Gastric or Duodenal Hemorrhagic Lesion
Description: Summary of data on the presence or absence of gastric or duodenal hemorrhagic lesion.
Time Frame: From baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3248
participants
  No | 3244
  Yes | 4

5. Secondary Outcome: Presence of Either Gastric/Duodenal Ulcer, or Gastric/Duodenal Hemorrhagic Lesion
Description: Summary of data on the presence or absence of gastric/duodenal ulcer gastric/duodenal hemorrhagic lesion.
Time Frame: From baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3248
participants
  No | 3237
  Yes | 11

6. Secondary Outcome: Treatment for Gastric/Duodenal Ulcer or Lesion
Description: Summary of data on the presence or absence of treatment for duodenal ulcers or hemorrhagic lesions.
Time Frame: From baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3248
participants
  No | 0
  Yes | 11

7. Secondary Outcome: Details of Treatment for Gastric or Duodenal Ulcers or Hemorrhagic Lesions
Description: Summary of data on the details of treatment for gastric or duodenal ulcers or hemorrhagic lesions.
  Participants could be counted in more than 1 treatment category.
Time Frame: From baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3248
participants
  Takepron Capsule or OD Tablets 15 mg | 4
  Takepron Capsule or OD Tablet 30 mg | 1
  Rabeprazole tablet 10 mg | 1
  Rabeprazole tablet 20 mg | 1
  H2 receptor antagonist (oral) | 1
  Other peptic ulcer medication | 4
  Endoscopic hemostasis | 1
  Other | 4

8. Secondary Outcome: Treatment Outcome (Including Duplicates) for Gastric or Duodenal Ulcers or Hemorrhagic Lesions
Description: Summary of data on the outcome of treatment for gastric or duodenal ulcers or hemorrhagic lesions.
Time Frame: From baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3248
participants
  Takepron 15 mg - Resolving | 3
  Takepron 15 mg - Unknown | 1
  Takepron 30 mg - Resolved | 1
  Rabeprazole 10 mg _Resolved | 1
  Rabeprazole 20 mg - Resolved | 1
  H2 receptor antagonist - Resolved | 1
  Other peptic ulcer medication - Resolved | 3
  Other peptic ulcer medication - Resolving | 1
  Endoscopic hemostasis - Resolving | 1
  Other - Resolved | 1
  Other - Resolving | 3

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. Among these, events which are considered possibly associated with a medicinal product are defined as adverse drug reactions.
Arm/Group | Lansoprazole 15 mg
Serious Adverse Events (participants affected / at risk) | 50/3302
Other Adverse Events (participants affected / at risk) | 0/3302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lansoprazole 15 mg (N=3302)
Cellulitis (Infections and infestations) | 2
Meningitis bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Delirium (Psychiatric disorders) | 1
Cerebral artery embolism (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Cervical myelopathy (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 3
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Bladder tamponade (Renal and urinary disorders) | 1
Malaise (General disorders) | 1
General physical health deterioration (General disorders) | 2
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Nephrectomy (Surgical and medical procedures) | 1
Incisional drainage (Surgical and medical procedures) | 1
Spinal operation (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.